CLINICAL TRIAL: NCT05387564
Title: Increasing Documentation and Disclosure of Sickle Cell Trait Status: An Implementation Science Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Corinna Schultz, Attending Physician, Nemours Children's Clinic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 348506
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Trait
Keywords: electronic health record; pediatric; newborn screen; implementation
MeSH Terms: conditions — Sickle Cell Trait

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "All-in" (Active Comparator): In the "all-in" arm, pediatric primary care physicians receive all toolkit components at once.
  Interventions: Behavioral: SCT Documentation and Disclosure Toolkit (SCT-DD)
- "Add-in" (Active Comparator): In the "add-in" arm, pediatric primary care physicians will have sequential addition of toolkit components in 6 week increments
  Interventions: Behavioral: SCT Documentation and Disclosure Toolkit (SCT-DD)

INTERVENTIONS:
Behavioral: SCT Documentation and Disclosure Toolkit (SCT-DD) — A toolkit of implementation strategies

SUMMARY:
The hemoglobinopathy newborn screen (NBS) performed on all neonates in the U.S. allows for early life-saving medical care for infants with sickle cell disease (SCD), an autosomal recessive genetic disorder. Because of its detection method, the NBS incidentally reveals hemoglobinopathy traits including sickle cell trait (SCT). In an effort to uphold the rights of the newborn to their medical data and preserve autonomy in medical decision making, pediatric and genetic society guidelines recommend disclosure and documentation of SCT results during infancy. Despite this guidance, a large guideline-to-practice gap exists: SCT status is grossly under-documented in the pediatric electronic health record and few adults report knowing their SCT status despite universal screening. We plan to evaluate the effect of a toolkit of SCT Documentation and Disclosure (SCT-DD) strategies on documentation and disclosure of SCT by pediatric primary care providers in a 2-arm randomized interrupted time series trial.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient pediatric primary care providers within Nemours and their patients

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Schultz, MD, MSHP, Principal Investigator — Nemours
Locations (1):
- Nemours Children's Hospital, Delware, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Invitations were sent to the "physician in charge" of 20 pediatric primary care sites within one hospital system in the mid-Atlantic region. Seven (7) sites were interested in participating in the pilot project and randomized to intervention arms. Clinicians and caregivers at each site were then recruited via email. Each group of participants is designated as a separate time period below: Clinicians, Caregivers from the retrospective period, caregivers from the prospective time.
Units Other Than Participants: Clinic Location
Period: Clinician
Arm/Group | "All-in" | "Add-in"
Started (Enrolled at Time point 0 (prior to intervention roll-out) and completed at least one survey) | 16; 4 Clinic Location | 12; 3 Clinic Location
Completed | 16; 4 Clinic Location | 12; 3 Clinic Location
Not Completed | 0; 0 Clinic Location | 0; 0 Clinic Location
Period: Caregiver Survey From Retrospective Time
Arm/Group | "All-in" | "Add-in"
Started (Number of Caregivers who consented to fill out a survey during the "retrospective" period before interventions rolled out to offices) | 22; 4 Clinic Location | 22; 3 Clinic Location
Completed (Number of Caregivers who filled out a survey during the "retrospective" period before interventions rolled out to offices) | 22; 4 Clinic Location | 22; 3 Clinic Location
Not Completed | 0; 0 Clinic Location | 0; 0 Clinic Location
Period: Caregiver Survey From Intervention Time
Arm/Group | "All-in" | "Add-in"
Started (Number of Caregivers who consented to fill out a survey during the "Intervention" period after interventions rolled out to offices) | 15; 4 Clinic Location | 27; 3 Clinic Location
Completed (Number of Caregivers who filled out a survey during the "Intervention" period after interventions rolled out to offices) | 15; 4 Clinic Location | 27; 3 Clinic Location
Not Completed | 0; 0 Clinic Location | 0; 0 Clinic Location

BASELINE CHARACTERISTICS:
Population: Two sets of participants included: 1) Physicians who were the primary target of the intervention, 2) Caregivers who consented and completed surveys. As physicians were the primary interest, demographic characteristics and the majority of study outcomes were based on physicians enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | "All-in" | "Add-in" | Total
Number analyzed (Participants) | 53 | 61 | 114
Age, Categorical [Count of Participants; unit: Participants] — Two sets of participants included: 1) Physicians who were the primary target of the intervention, 2) Caregivers who consented and completed surveys. As physicians were the primary interest, demographic characteristics and the majority of study outcomes were based on physicians enrolled. Population: Physician population only
  Participants
    number analyzed (Participants) | 16 | 12 | 28
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 16 | 12 | 28
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two sets of participants included: 1) Physicians who were the primary target of the intervention, 2) Caregivers who consented and completed surveys. As physicians were the primary interest, demographic characteristics and the majority of study outcomes were based on physicians enrolled.
  Participants
    Physicians: number analyzed (Participants) | 16 | 12 | 28
    Physicians: Female | 13 | 8 | 21
    Physicians: Male | 3 | 4 | 7
    Caregivers who completed surveys: number analyzed (Participants) | 37 | 49 | 86
    Caregivers who completed surveys: Female | 36 | 49 | 85
    Caregivers who completed surveys: Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race/Ethnicity not collected from Caregiver Survey Participants Population: Two sets of participants included: 1) Physicians who were the primary target of the intervention, 2) Caregivers who consented and completed surveys. As physicians were the primary interest, demographic characteristics and the majority of study outcomes were based on physicians enrolled.
  Participants
    Physicians: number analyzed (Participants) | 16 | 12 | 28
    Physicians: American Indian or Alaska Native | 0 | 0 | 0
    Physicians: Asian | 2 | 2 | 4
    Physicians: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Physicians: Black or African American | 0 | 2 | 2
    Physicians: White | 13 | 8 | 21
    Physicians: More than one race | 0 | 0 | 0
    Physicians: Unknown or Not Reported | 1 | 0 | 1
    Caregivers who completed surveys: number analyzed (Participants) | 37 | 49 | 86
    Caregivers who completed surveys: American Indian or Alaska Native | 1 | 1 | 2
    Caregivers who completed surveys: Asian | 2 | 1 | 3
    Caregivers who completed surveys: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers who completed surveys: Black or African American | 8 | 27 | 35
    Caregivers who completed surveys: White | 21 | 17 | 38
    Caregivers who completed surveys: More than one race | 2 | 1 | 3
    Caregivers who completed surveys: Unknown or Not Reported | 3 | 2 | 5
Confidence regarding hemoglobinopathies [Mean (Standard Deviation); unit: units on a scale (1-10, 10 'extremely')] — On-line survey of confidence regarding the hemoglobinopathy newborn screen. Scale of 1-10. (1, least confident. 10, most confident). Population: Based on physicians enrolled (not caregivers)
  units on a scale (1-10, 10 'extremely')
    Confidence to interpret the hemoglobinopathy newborn screen results: number analyzed (Participants) | 16 | 12 | 28
    Confidence to interpret the hemoglobinopathy newborn screen results | 7.33 (2.2) | 7.33 (2.0) | 7.33 (2.1)
    Confidence to discuss hemoglobinopathy results with family: number analyzed (Participants) | 16 | 12 | 28
    Confidence to discuss hemoglobinopathy results with family | 8.08 (1.83) | 7.5 (1.7) | 7.75 (1.76)
    Confidence to discuss inheritance of hemoglobinopathies: number analyzed (Participants) | 16 | 12 | 28
    Confidence to discuss inheritance of hemoglobinopathies | 7.19 (2.07) | 8.50 (2.20) | 7.75 (2.19)
    Confidence to discuss reproductive options for hemoglobinopathies: number analyzed (Participants) | 16 | 12 | 28
    Confidence to discuss reproductive options for hemoglobinopathies | 5.8 (2.21) | 6.25 (2.99) | 6.00 (2.54)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: Acceptability of toolkit components by pediatric primary care providers by survey at the end of the study (i.e. 18 weeks after initial roll-out of interventions). Reported as the number who answered Agree or Strongly Agree on a 4-point Likert scale that they liked the toolkit component. Likert scale options included strong disagree, disagree, agree, strongly agree.
Time Frame: At conclusion of study: 18 weeks after initial roll-out of interventions
Population: At conclusion of study: 18 weeks after initial roll-out of interventions.
Measure: Count of Participants; unit: Participants
Arm/Group | "All-in" | "Add-in"
Number analyzed (Participants) | 13 | 10
Participants
  Liked the newborn screen EPIC prompt | 11 | 8
  Liked the educational module | 11 | 8
  Liked the reference materials | 10 | 5

2. Primary Outcome: Self-efficacy
Description: Confidence to document/discuss SCT result by pediatric primary care providers by survey. Scale 1 to 10: 1 = not confident at all, 10 = extremely confident.
Time Frame: At conclusion of study (18 weeks after initial roll-out of interventions)
Population: Based on participants who answered final survey at 18 weeks post intervention
Measure: Mean (Standard Deviation); unit: units on a scale (1-10)
Arm/Group | "All-in" | "Add-in"
Number analyzed (Participants) | 16 | 12
units on a scale (1-10)
  Confidence to interpret the hemoglobinopathy newborn screen results: number analyzed (Participants) | 13 | 10
  Confidence to interpret the hemoglobinopathy newborn screen results | 8.55 (1.37) | 8.20 (1.32)
  Confidence to discuss hemoglobinopathy results: number analyzed (Participants) | 13 | 10
  Confidence to discuss hemoglobinopathy results | 8.27 (1.35) | 8.8 (0.78)
  Confidence to discuss inheritance of hemoglobinopathies: number analyzed (Participants) | 13 | 10
  Confidence to discuss inheritance of hemoglobinopathies | 8.73 (1.42) | 8.89 (0.92)
  Confidence to discuss reproductive options of hemoglobinopathies: number analyzed (Participants) | 13 | 10
  Confidence to discuss reproductive options of hemoglobinopathies | 6.18 (2.48) | 7.0 (2.36)

3. Primary Outcome: Feasibility of Using Toolkit Components
Description: Number of pediatric primary care providers who used individual toolkit components in the last 6 weeks of the study (week 12-18) as indicated by answering "yes" to questions about whether individual toolkit components were used on a survey at the end of the study (18 weeks after roll-out of interventions).
Time Frame: Survey at end of study: 18 weeks after roll-out of interventions
Measure: Count of Participants; unit: Participants
Arm/Group | "All-in" | "Add-in"
Number analyzed (Participants) | 16 | 12
Participants
  EHR Prompt | 13 | 10
  Educational video | 12 | 9
  Reference Materials | 11 | 8

4. Secondary Outcome: Knowledge
Description: Knowledge of newborn screen results by caregivers via survey.
Time Frame: Survey for retrospective patients was sent before intervention roll-out. Survey for prospective patients were sent on a rolling basis at 2 months of age for any newborn patient seen during the 18 week intervention period.
Population: Surveys completed
Measure: Count of Participants; unit: Participants
Groups:
- "All-in": In the "all-in" arm, pediatric primary care physicians received all toolkit components at once.
Arm/Group | "All-in" | "Add-in"
Number analyzed (Participants) | 37 | 49
Participants
  Survey respondents who reported they received newborn screen results - Retrospective: number analyzed (Participants) | 22 | 22
  Survey respondents who reported they received newborn screen results - Retrospective | 14 | 15
  Survey respondents who reported they received newborn screen results - Prospective: number analyzed (Participants) | 15 | 27
  Survey respondents who reported they received newborn screen results - Prospective | 6 | 18
  Survey respondents who reported sickle cell trait on their child's newborn screen -Retrospective: number analyzed (Participants) | 22 | 22
  Survey respondents who reported sickle cell trait on their child's newborn screen -Retrospective | 0 | 2
  Survey respondents who reported sickle cell trait on their child's newborn screen -Prospective: number analyzed (Participants) | 15 | 27
  Survey respondents who reported sickle cell trait on their child's newborn screen -Prospective | 0 | 1

5. Primary Outcome: Penetration
Description: The number of newborns with newborn screen results visible in the electronic healthcare record and presence of documentation of abnormal newborn screen results. By chart review.
Time Frame: Chart review for retrospective patients was done before intervention roll-out. Chart review for prospective patients was done on a rolling basis at 2 months of age for any newborn patient seen during the 18 week intervention period
Population: Number of newborn patients in the all-in and add-in arms who were seen at sites enrolled in the trial during the retrospective and prospective periods. Chart reviews completed on all patients. Chart review for retrospective patients was done before intervention roll-out. Chart review for prospective patients was done at 2 months of age.
Measure: Count of Participants; unit: Participants
Groups:
- "Add in": In the "add-in" arm, pediatric primary care physicians received toolkit components in 6 week increments.
Arm/Group | "All-in" | "Add in"
Number analyzed (Participants) | 881 | 825
Participants
  Newborn screen available in EPIC - Retrospective: number analyzed (Participants) | 625 | 534
  Newborn screen available in EPIC - Retrospective | 424 | 303
  Newborn screen available in Careeverywhere - Retrospective: number analyzed (Participants) | 625 | 534
  Newborn screen available in Careeverywhere - Retrospective | 167 | 179
  Sickle cell trait on newborn screen - Retrospective: number analyzed (Participants) | 625 | 534
  Sickle cell trait on newborn screen - Retrospective | 9 | 13
  Sickle cell trait on problem list - Retrospective: number analyzed (Participants) | 625 | 534
  Sickle cell trait on problem list - Retrospective | 4 | 11
  Sickle cell trait documented as disclosed - Retrospective: number analyzed (Participants) | 625 | 534
  Sickle cell trait documented as disclosed - Retrospective | 4 | 2
  Newborn screen available in EPIC - Prospective: number analyzed (Participants) | 256 | 291
  Newborn screen available in EPIC - Prospective | 190 | 190
  Newborn screen available in Careeverywhere - Prospective: number analyzed (Participants) | 256 | 291
  Newborn screen available in Careeverywhere - Prospective | 54 | 70
  Sickle cell trait on newborn screen - Prospective: number analyzed (Participants) | 256 | 291
  Sickle cell trait on newborn screen - Prospective | 4 | 9
  Sickle cell trait on problem list - Prospective: number analyzed (Participants) | 256 | 291
  Sickle cell trait on problem list - Prospective | 3 | 9
  Sickle cell trait documented as disclosed - Prospective: number analyzed (Participants) | 256 | 291
  Sickle cell trait documented as disclosed - Prospective | 3 | 4

ADVERSE EVENTS:
Time Frame: For Physicians: From enrollment until last survey completed (total 18 weeks). Adverse events not evaluated from chart review or caregiver surveys
Arm/Group | "All-in" | "Add-in"
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 0/16 | 0/12

LIMITATIONS AND CAVEATS:
Very small number of caregivers of children with sickle cell trait responded to survey requests.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT05387564/Prot_SAP_000.pdf